CLINICAL TRIAL: NCT06305364
Title: Predicting Adenomatous Polyps in the Colon, Using Images of a Human Tongue
Brief Title: Predicting Adenomatous Polyps in the Colon Using Images of a Human Tongue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jubaan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL-1001
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Neoplasms; Gastrointestinal Microbiome
Keywords: Artificial Intelligence
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Masking Description: Gastroenterologist performing standard of care colonoscopy post Gixam test will be blinded to the Gixam prediction score.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Gixam followed by standard of care colonoscopy (Experimental): This is a single-arm study. All participants will undergo the Gixam test following a standard of care colonoscopy
  Interventions: Device: Gixam

INTERVENTIONS:
Device: Gixam — Participants will be required to extend their tongue in the Gixam device. Six images will be obtained and analyzed by the artificial intelligence (AI) model generating a prediction score for the presence of colorectal adenoma.

SUMMARY:
This is a prospective, multicenter, single-arm clinical investigation designed to evaluate the accuracy of the Gixam™ System in identifying subjects with colorectal adenomas compared to optical colonoscopy. Subjects arriving for a standard of care colonoscopy at the investigation site will be offered to participate in the study. Following an informed consent process, images of the subjects' tongue will be obtained with the Gixam™ System and a prediction score will be generated by the Gixam™ AI model. Subjects will thereafter proceed to their SOC colonoscopy, and the Gixam™ score will be compare with colonoscopy findings to evaluate its performance.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females
2. Age: 18-75 years, inclusive
3. Scheduled for colonoscopy procedure at investigation site subject to one of the below criteria:

   1. Screening - defined as first colonoscopy or consecutive colonoscopy without previous findings, previous colonoscopy performed at least 10 years ago (- 1 year);
   2. Patient with finding of colorectal adenoma or sessile serrated polyp in previous colonoscopy (must be documented in patient's medical history).
4. Able to comprehend and provide informed consent.

Exclusion Criteria:

1. Subject who is not a suitable candidate for a colonoscopy
2. Lynch or Familial Adenomatous Polyposis (FAP) inherited syndromes
3. Current or previous Inflammatory Bowel Disease (IBD - Crohn's, Ulcerative Colitis) of significant duration
4. Patients with a disability to extend their tongue.
5. Patients with tongue piercings.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Number of device related adverse events and serious adverse events | 1 day
Primary Efficacy Endpoint - Gixam's diagnostic accuracy | 14 days (till pathology report is received)
  Gixam's diagnostic accuracy (sensitivity and specificity) of adenomatous colorectal polyps.
  The Gixam's predictive value will be compared to the patient's colonoscopy + pathology (if any specimens are collected) findings as ground truth on a binary basis (YES/NO for adenomatous and sessile serrated polyps).

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Bleistein, Study Director — Jubaan Ltd.
Locations (3):
- United States (3):
  - NYU Langone Health, New York, New York
  - Westside GI, New York, New York
  - NewYork-Presbyterian / Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jubaan's website — https://jubaan.com/